CLINICAL TRIAL: NCT04578210
Title: A Phase I/II Dose-escalation Multi Center Study to Evaluate the Safety of Infusion of NatuRal KillEr celLs or MEmory T Cells as Adoptive Therapy in coronaviruS pnEumonia and/or Lymphopenia
Brief Title: Safety Infusion of NatuRal KillEr celLs or MEmory T Cells as Adoptive Therapy in COVID-19 pnEumonia or Lymphopenia
Acronym: RELEASE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Universidad Autonoma de Madrid (Other); Universidad Miguel Hernandez de Elche (Other); Biobizkaia Health Research Institute (Other Government); Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RELEASE
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2022-05

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Phase I/II escalating-dose clinical trial, randomized study to determine safety, tolerability, alloreactivity and efficacy of cell therapy with adoptive cell therapy of NK cells or memory T cells in patients affected by COVID-19 Donors will be patients recovered from COVID-19 Will be 2 arms
  * A: allogeneic T memory cells
  * B: allogeneic NK cells
  Two consecutive phases:
  * The first dose escalation focuses on determining safety and the recommended dose for the phase II Phase I: Patients with SARS-CoV-2+ pneumonia and/or lymphopenia and O2Sat ≤ 94% on room air at screening, with no oxygen required or with an oxygen need of ≤ 2.5 lpm in nasal cannula, will be selected This phase has a single ascending dose design with up to 3 planned dose levels for each arm.
  * The second phase extends the safety study Phase II: Patients with SARS-CoV-2+ pneumonia and/or lymphopenia and O2Sat ≤ 94% on room air at screening, requiring or not oxygen supplementation
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: allogeneic T memory cells (Experimental): patients will receive memory T cells
  Interventions: Biological: T memory cells and NK cells
- Arm B: allogeneic NK cells (Experimental): patients will receive NK cells
  Interventions: Biological: T memory cells and NK cells

INTERVENTIONS:
Biological: T memory cells and NK cells — Single infusion of NK or memory T cells from a healthy donor recovered from COVID-19 (dose escalation).

SUMMARY:
This is a phase I/II clinical trial using adoptive cell therapy with NK cells or memory T cells in patients affected by COVID-19.

Severe cases with COVID-19 present a dysregulated immune system with T cell lymphopenia, specially NK cells and memory T cells, and a hyper-inflammatory state.

This clinical trial proposes the use of cell therapy for the treatment of patients with worse prognosis due to SARS-CoV-2 infection (those with pneumonia and/or lymphopenia). This is an innovative and a non-pharmacological intervention.

DETAILED DESCRIPTION:
In this phase I/II trial natural killer (NK) cells or memory T lymphocytes will be infused from donors who have recovered from COVID-19 and have complete resolution of symptoms for at least 14 days.

There will be two arms based on the biology of the donor and the patient:

Arm 1. Infusion of memory T cells from HLA partially match donors which have the SARS-COV-2 memory T cell repertoire.

Arm 2. Infusion of NK cells which are cells of the innate immune system that can eliminate virally infected cells.

The investigators expect a quick recovery of the patients with pneumonia or lymphopenia for two reasons:

1. The pool of memory T cells will increase in patients. Memory T cell levels are low in these patients. These lymphocytes have long-life memory, which upon reencountering SARS-CoV-2 will induce enhanced effector function resulting in greater protection of the patient.
2. NK cells act quickly after a viral infection. The number and function of NK cells correlates with the severity of another coronavirus infection, Severe Acute Respiratory Syndrome (SARS), originated in China in 2002.

Moreover, the investigators have previous successful experience with other viruses such as CMV, EBV and HHV-6.

Patients who have recovered from COVID-19 are the ideal donor candidates because they have immune cells with memory against SARS-CoV-2. Therefore, the infusion of NK and memory T cells from these donors will increase the pool of cells with cytotoxicity to virally infected cells, and will increase the pool of memory cells that respond quicker to a previously encountered stimulus.

This will impact in saving thousands of lives, releasing hospital beds, reducing the costs of a national health system and improving the economy of a locked-down country.

Cell therapies are safe and cost-effective and successfully used in other diseases. The investigators need new innovative treatments where others have failed.

We have performed the phase I:

Arm 1.Phase I single-center dose-escalation in 9 patients infused with memory T cells from a HLA partially match convalescent donor.

Arm 2. Phase I single-center dose-escalation in 6 patients infused with NK cells from convalescent donors.

We evaluate the safety, and feasibility, and obtained the RP2D of a single infusion.

We have performed the phase II with memory T cells:

The phase II for the infusion of memory T cells from HLA partially match convalescent donors has been carried out. 84 patients have been enrolled and randomized into the SoC treatment or the SoC plus the infusion of memory T cells.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≤ 80 years of age.
* Patient with diagnosis of COVID-19 infection with laboratory confirmation by reverse-transcription PCR (RT-PCR) of SARS-CoV-2 <72 hours prior to study entry.
* Onset of symptoms < 10 days prior to administration of study treatment.
* No more than 72 hours (3 days) of hospitalization before study treatment administration.
* Phase I criteria: Patients requiring hospitalization for COVID-19, with pneumonia diagnosed with chest radiograph or computed tomography imaging or lymphopenia (absolute lymphocyte counts below 1.2 x 109cells /L) AND O2Sat ≤ 94% on room air at screening, no oxygen requirement or with an oxygen need of ≤ 2.5 lpm in nasal cannula.
* Phase II criteria: Patients requiring hospitalization with pneumonia diagnosed with chest radiograph or computed tomography imaging or lymphopenia (absolute lymphocyte counts below 1.2 x 109cells /L) AND O2Sat ≤ 94% on room air at screening, requiring or not oxygen supplementation (nasal cannula, oxygen mask with reservoir, non-invasive ventilation, etc), but excluding mechanical ventilation.
* Have a negative pregnancy test documented prior to enrollment (for females of childbearing potential).
* Be willing and able to comply with study procedures.
* Patients with the ability to comprehend and sign the informed consent
* Written informed consent obtained prior to any screening procedures.

Exclusion Criteria:

* Enrolled in another Clinical Trial for COVID19.
* Rapidly progressive disease with anticipated life-expectancy <72 hours.
* Patients requiring mechanical ventilation.
* Patients with multiorgan failure.
* Mild-moderate (grade ≥ 3) organ impairment (liver, kidney, respiratory), according to criteria from the National Cancer Institute (NCI CTCAE version 5.0).
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol.
* Have a known history of human immunodeficiency virus infection, Hepatitis B or Hepatitis C; testing is not required in the absence of prior documentation or known history.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Any other condition that, in the opinion if the Investigator, may interfere with the efficacy and/or safety evaluation of the trial.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Phase I: Occurrence of DLTs in all patients during the study treatment, until 21 days after cell infusion and the MTD | 3 months
  Any grade 3 or higher toxicity with an attribution of definitely or probably related to the infusion of the cells and any lower grade toxicity that increases to a grade 3 or higher as a direct result of the cell infusion.
Phase II | 3 months
  Phase II primary outcome is the incidence of patient recovery infusing adoptive NK cells or adoptive memory T cells. Recovery is defined as the proportion of participants in each group with normalization of fever and oxygen saturation (criteria for normalization: temperature < 38°C armpit, and SpO2 > 94%, sustained for at least 24 h) or lymphopenia recovery through day 14.

SECONDARY OUTCOMES:
Secondary Outcomes | 3 months
  Time (days) to normal level of lymphocytes. Proportion of patients showing clinical improvement at day 7 according to the investigator (based on respiratory status and blood-result tests).
  Proportion of patients receiving a second cycle. Time (days) to first negative SARS-CoV-2 PCR after infusing adoptive NK cells or adoptive memory T cells.
  The incidence of treatment-related adverse events (new or worsening from baseline) Duration (days) of hospitalization. Time (days) to discharge or to a NEWS of ≤ 2 and maintained for 24 hours, whichever comes first.
  Time to improvement by one category on a 7-point ordinal scale. Subject clinical status (on a 7-point ordinal scale) at day 14. Proportion of patients requiring intensive care unit. All-cause mortality at Day 28.

OTHER OUTCOMES:
Exploratory Outcomes | 3 months
  To determine donor chimerism by short tandem repeats and a variable number of tandem repeat markers using the ABI Prism 3130 System and immune lymphocyte reconstitution by multiparametric flow cytometry after adoptive therapy weekly during the first month after infusion.
  Immune reconstitution: Immunoglobulins, serum cytokines (IL-6, IL-1, TNFa, IFNb, IL-10); T cell repertoire: CD3 (CD4, CD8), naive CD45RA+CD27+, central memory CD45RA-CD27+, effector memory CD45RA-CD27- y EMRA CD45RA+CD27-, Activated T cells (HLADR+), T regs (CD4+CD25+CD127low), Tgd; NK cells repertoire CD56+CD3- (KIR (2DL1, 2DL2/3, 3DL1), NCR (NKp30, NKp44, NKp46), NKG2D); NKT cells, B cells, memory B cells (CD19+CD27+).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferreras C, Hernandez-Blanco C, Martin-Quiros A, Al-Akioui-Sanz K, Mora-Rillo M, Ibanez F, Diaz-Almiron M, Cano-Ochando J, Lozano-Ojalvo D, Jimenez-Gonzalez M, Goterris R, Sanchez-Zapardiel E, de Paz R, Guerra-Garcia P, Queiruga-Parada J, Molina P, Briones ML, Ruz-Caracuel B, Borobia AM, Carcas AJ, Planelles D, Vicario JL, Moreno MA, Balas A, Llano M, Llorente A, Del Balzo A, Canada C, Garcia MA, Calvin ME, Arenas I, Perez de Diego R, Eguizabal C, Soria B, Solano C, Perez-Martinez A. Results of phase 2 randomized multi-center study to evaluate the safety and efficacy of infusion of memory T cells as adoptive therapy in severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pneumonia and/or lymphopenia (RELEASE NCT04578210). Cytotherapy. 2024 Jan;26(1):25-35. doi: 10.1016/j.jcyt.2023.10.002. Epub 2023 Oct 29. PMID 37897472
- [Derived] Herrera L, Martin-Inaraja M, Santos S, Ingles-Ferrandiz M, Azkarate A, Perez-Vaquero MA, Vesga MA, Vicario JL, Soria B, Solano C, De Paz R, Marcos A, Ferreras C, Perez-Martinez A, Eguizabal C. Identifying SARS-CoV-2 'memory' NK cells from COVID-19 convalescent donors for adoptive cell therapy. Immunology. 2022 Feb;165(2):234-249. doi: 10.1111/imm.13432. Epub 2021 Dec 2. PMID 34775592
- [Derived] Garcia-Garcia I, Guerra-Garcia P, Ferreras C, Borobia AM, Carcas AJ, Queiruga-Parada J, Vicario JL, Mirones I, Solano C, Eguizabal C, Soria B, Perez-Martinez A. A phase I/II dose-escalation multi-center study to evaluate the safety of infusion of natural killer cells or memory T cells as adoptive therapy in coronavirus pneumonia and/or lymphopenia: RELEASE study protocol. Trials. 2021 Oct 2;22(1):674. doi: 10.1186/s13063-021-05625-7. PMID 34600562
- [Derived] Perez-Martinez A, Mora-Rillo M, Ferreras C, Guerra-Garcia P, Pascual-Miguel B, Mestre-Duran C, Borobia AM, Carcas AJ, Queiruga-Parada J, Garcia I, Sanchez-Zapardiel E, Gasior M, De Paz R, Marcos A, Vicario JL, Balas A, Moreno MA, Eguizabal C, Solano C, Arribas JR, Buckley RM, Montejano R, Soria B. Phase I dose-escalation single centre clinical trial to evaluate the safety of infusion of memory T cells as adoptive therapy in COVID-19 (RELEASE). EClinicalMedicine. 2021 Sep;39:101086. doi: 10.1016/j.eclinm.2021.101086. Epub 2021 Aug 13. PMID 34405140
- [Derived] Del Pozo Martin Y. 47th Annual Meeting of the EBMT. Lancet Haematol. 2021 May;8(5):e317-e318. doi: 10.1016/S2352-3026(21)00104-6. Epub 2021 Mar 31. No abstract available. PMID 33811823